CLINICAL TRIAL: NCT05418816
Title: Initial Feasibility Study of SelfWrap-Assisted Arteriovenous Fistulas (SW-AVF)
Brief Title: SelfWrap-Assisted Arteriovenous Fistulas
Acronym: SW-AVF
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VenoStent (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PLN-030
Record Dates: First submitted 2022-06-07; First posted 2022-06-14 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Chronic Kidney Diseases; Chronic Kidney Failure; End Stage Renal Disease; End Stage Kidney Disease; Arteriovenous Fistula; Hemodialysis Access Failure; Catheter Complications; Catheter Dysfunction; Vascular Diseases; Arteriovenous Malformations; Vascular Malformations; Vascular Fistula; Fistula; Renal Insufficiency; Renal Failure; Renal Failure Chronic; Urologic Diseases
Keywords: Dialysis; Hemodialysis; Chronic Kidney Disease; End Stage Renal Disease; Vascular Surgery; Vascular Access; Arteriovenous Fistula; AVF; Nephrology; Bioabsorbable; Perivascular Wrap; External Support
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic; Arteriovenous Fistula; Vascular Diseases; Arteriovenous Malformations; Vascular Malformations; Vascular Fistula; Fistula; Renal Insufficiency; Urologic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- SelfWrap-treated (Experimental): Treated with SelfWrap Bioabsorbable Perivascular Wrap during AVF creation surgery
  Interventions: Device: SelfWrap Bioabsorbable Perivascular Wrap

INTERVENTIONS:
Device: SelfWrap Bioabsorbable Perivascular Wrap — SelfWrap is applied during the normal arteriovenous fistula (AVF) creation procedure. It provides mechanical support to the vein and induces outward remodeling to improve maturation and patency of AVFs.
  Other Names: SelfWrap

SUMMARY:
This is a single-center, prospective, single-arm clinical study to evaluate the feasibility, safety, and performance of VenoStent's SelfWrap® Bioabsorbable Perivascular Wrap on arteriovenous fistulas (AVFs). All participants are chronic kidney disease (CKD) patients already receiving hemodialysis treatments that are referred for creation of a new arteriovenous fistula (AVF).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years, male or female;
2. Subjects already receiving hemodialysis treatments that are ultimately referred for a new AVF, per current US KDOQI Clinical Practice Guidelines for Vascular Access updated in 2019 which recommend an AVF or arteriovenous graft (AVG) consistent with patient life-plan, overall goals of care, and anticipated duration of hemodialysis; if life expectancy > 1 year, recommend forearm AVF, forearm AVG, or upper arm AVF; if < 1 year, recommend forearm AVG/upper arm AVG; if urgent start, early cannulation AVG or central venous catheter (CVC);
3. Target cephalic vein inner diameter ≥ 2.5 mm and target artery ≥ 2.0 mm as measured via duplex ultrasound with a tourniquet applied;
4. For radial AVFs, a nonpathological modified Allen test;
5. Triphasic arterial flow and intact venous outflow;
6. A vascular access site being used for hemodialysis that is either positioned contralateral to the planned AVF creation surgery or located in the groin. If the catheter is positioned on the same side as the planned AVF, the catheter will be moved to the other arm prior to the AVF created surgery.
7. Participant is willing and able to comply with study requirements and sign an informed consent.

Exclusion Criteria:

1. Planned index procedure to revise or repair an existing fistula;
2. Twelve months or longer with a catheter, on the planned side of AVF creation; or if there has been any previously failed AVF and AVG on the planned side of AVF creation.
3. Significant (> 50%) stenosis at the target vein on the side of surgery, as diagnosed by preoperative ultrasound;
4. Known central venous stenosis > 50%;
5. Amputated limb;
6. Use of a peripherally-inserted central catheter (PICC) line;
7. Abnormal cardiac rhythm;
8. Known coagulation disorder;
9. Known or suspected active infection at the time of surgery;
10. Congestive heart failure NYHA class 4;
11. Prior steal on the side of surgery;
12. Enrolled in another investigational drug, device, or biological study and has not completed the primary endpoint(s), or was previously enrolled in this study;
13. Life expectancy less than 12 months;
14. Patient expecting to undergo kidney transplant surgery within 12 months of enrollment;
15. Patient has a comorbid condition that, in the judgment of the Investigator, may cause him/her to be non-compliant with the protocol or confound data interpretation.
16. Unwillingness or inability to give consent and/or comply with the study follow up schedule.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-06-14 (Actual); Primary Completion 2022-02-23 (Actual); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Primary Patency | Through 6 months post-AVF creation
  Proportion of participants with a created AVF that is not abandoned nor occluded and is free from access thrombosis as well as any intervention required to facilitate, maintain, or reestablish patency (e.g. angioplasty), through 6 months
Cumulative Patency | Through 6 months post-AVF creation
  Proportion of participants with a created AVF that is not abandoned or occluded, through 6 months
Freedom from Device-Related Safety Events | Through 6 months post-AVF creation
  Proportion of participants with freedom from device-related infection, thrombosis, aneurysm, pseudoaneurysm, major bleeding, and rehospitalizations

SECONDARY OUTCOMES:
Primary Patency | Through 1, 2, 3, 12, 18, and 24 months post-AVF creation
  Proportion of participants with a created AVF that is not abandoned nor occluded and is free from access thrombosis as well as any intervention required to facilitate, maintain, or reestablish patency (e.g. angioplasty), through 1, 2, 3, and 12 months
Cumulative Patency | Through 1, 2, 3, 12, 18, and 24 months post-AVF creation
  Proportion of participants with a created AVF that is not abandoned or occluded, through 1, 2, 3, and 12 months
Number of Interventions | Through 1, 2, 3, 6, 12, 18, and 24 months post-AVF creation
Unassisted Physiological Maturation | 1, 2, 3, and 6 months post-AVF creation
  A created AVF with a proximal arterial flow rate ≥ 500 mL/min and a vein inner diameter ≥ 4.0 mm near the cannulation site, in absence of intervention(s) to initially establish this flow rate and vein size
Freedom from Device-Related Safety Events | Through 1, 2, 3, 12, 18, and 24 months post-AVF creation
  Proportion of participants with freedom from device-related infection, thrombosis, aneurysm, pseudoaneurysm, major bleeding, and rehospitalizations

OTHER OUTCOMES:
Assisted Physiological Maturation | 1, 2, 3, and 6 months post-AVF creation
  A created AVF with a proximal arterial flow rate ≥ 500 mL/min and a vein inner diameter ≥ 4.0 mm near the cannulation site, which required intervention(s) (e.g. angioplasty) to initially establish this flow rate and vein size
Assisted Primary Patency | 1, 2, 3, 6, 12, 18, and 24 months post-AVF creation
  Proportion of participants with a created AVF that is not abandoned nor occluded and is free from access thrombosis, through 1, 2, 3, 6, and 12 months
Time-to-Cannulation (or Cumulative Incidence) | Through 12 months
  The time from AVF creation to the first two-needle hemodialysis through the newly-created AVF, as reported by the clinical research associate or site-designated clinician
Time-to-Maturation (Functional Maturation) | Through 12 months
  The duration of time from AVF creation to the first date that the AVF is able to provide prescribed dialysis consistently with two needles for more than two thirds of dialysis sessions within 4 consecutive weeks, as reported by the CRA or site-designated clinician
Functional Primary Patency | 2, 3, 6, 12, 18, and 24 months
  Proportion of participants with a created AVF that is free from thrombosis as well as any intervention required to facilitate, maintain, or reestablish patency (e.g. angioplasty), from the first date that it is able to provide prescribed dialysis consistently with two needles for more than two thirds of dialysis sessions within 4 consecutive weeks (i.e. mature AVF) as reported by the CRA or site-designated clinician, at 2, 3, 6, and 12 months
Functional Cumulative Patency | 2, 3, 6, 12, 18, and 24 months
  Proportion of participants with a created AVF that is not abandoned or occluded, from the first date that it is able to provide prescribed dialysis consistently with two needles for more than two thirds of dialysis sessions within 4 consecutive weeks as reported by the CRA or site-designated clinician, at 2, 3, 6, and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Ebner, MD, Principal Investigator — Sanatorio Italiano
Locations (1):
- Sanatorio Italiano, Asunción, Paraguay

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: VenoStent website — https://www.venostent.com